CLINICAL TRIAL: NCT01353521
Title: Contrast-enhanced Ultrasound for the Evaluation of Complex Renal Cysts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Anil Kapoor, MD, FRCSC, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEUSEVCRC
Record Dates: First submitted 2011-03-11; First posted 2011-05-13 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Complex Renal Cyst
Keywords: complex renal cysts; Contrast enhanced ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast-enhanced ultrasound (Experimental)
  Interventions: Procedure: Contrast-enhanced ultrasound

INTERVENTIONS:
Procedure: Contrast-enhanced ultrasound — A contrast-enhanced ultrasound utilizes intravenous gas-filled microbubbles to enhance visualization in real time.
  Other Names: CEUS

SUMMARY:
Complex renal cysts are often incidentally detected on imaging. The differential diagnosis of the complex renal cyst includes various benign cystic lesions, which are based on the Bosniak classification scheme. Currently the standard of care in evaluating a complex renal cyst is using a contrast-enhanced computed tomography (CT) scan, or a contrast-enhanced magnetic resonance imaging (MRI) scan. Since both of these modalities present adverse events due to frequent high doses of radiation, a technique such as a contrast-enhanced ultrasound (CEUS) can be used to obtain the same results, without having to impose high doses of radiation upon a patient.

DETAILED DESCRIPTION:
By evaluating complex renal cysts using a contrast-enhanced ultrasound (CEUS), it can be established as to whether or not the results are better, the same, or worse, when compared to CT and/or MRI scans.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old and capable of giving informed consent
* all patients undergoing CT evaluation of complex renal cysts at our centre (either initially or in follow-up)
* A complex renal cyst defined as Bosniak IIF, III or IV

Exclusion Criteria:

* pregnant patients
* patients with contrast allergies
* patients with non-cystic, solid renal masses
* patients with simple cysts (Bosniak class I and II)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
concordance between CEUS and CT | (Baseline, follow up at 3, 6, 9, & 12 months)
  Complex renal cysts will be classified using the Bosniak classification system for both the CEUS and CT and compared. If surgical removal of a complex cyst is required (Bosniak IIF, III or IV), then the pathology will be evaluated with a single CEUS and a CT (The CEUS will be conducted 14 days within the CT).

SECONDARY OUTCOMES:
histopathological diagnosis after surgery of complex renal cysts | Baseline and every three months until the end of study.
Average percent difference of CEUS vs CT imaging | Baseline imaging (CEUS 14 days within a CT scan)
  If during watchful waiting another CEUS is needed to be done in cases where a CT scan does show change at a follow up visit, then this average percent difference will also be calculated at this point.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kapoor, MD, Principal Investigator — McMaster Institute of Urology - St. Joseph's Healthcare Hamilton; Christopher Allard, MD, Study Chair — McMaster Institute of Urology - St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada